CLINICAL TRIAL: NCT05864989
Title: Non-Incised Papilla Flap With and Without Connective Tissue Graft for Management of Deep Supraossous Defects
Brief Title: Non-Incised Papilla Flap in Deep Supraossous Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mahetab mohamed abdel el wahab, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1240
Record Dates: First submitted 2023-05-01; First posted 2023-05-18 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIPSA in deep supra-alveolar defects without connective tissue graft (Experimental)
  Interventions: Procedure: Non-incised papila surgical approach only
- NIPSA in deep supra-alveolar defects with connective tissue graft (Active Comparator)
  Interventions: Procedure: Non-incised papila surgical approach with connective tissue grafting

INTERVENTIONS:
Procedure: Non-incised papila surgical approach only — Reconstructive periodontal surgery
  Arms: NIPSA in deep supra-alveolar defects without connective tissue graft
Procedure: Non-incised papila surgical approach with connective tissue grafting — Reconstructive periodontal surgery
  Arms: NIPSA in deep supra-alveolar defects with connective tissue graft

SUMMARY:
The objective of this study was to assess the effectiveness of NIPSA in periodontal lesions with deep supra-alveolar defects, measuring the clinical efficacy of this flap. The non-incised papilla surgical approach (NIPSA) is a novel technique that accesses the periodontal defect from apical direction and was established with the aim of creating clinical advances compared with marginal access techniques.

The defects with a supra-alveolar components are more frequent than intrabony defects, there is very little evidence about their treatment .

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of periodontal disease (periodontitis stage III and IV, grade A [12];
* non-smokers and former smokers who quit smoking at least 1 year previously
* previous treatment for periodontal disease using non-surgical periodontal treatment completion of step I and II of periodontal therapy
* compliance with periodontal maintenance and oral hygiene (FMPS at baseline ≤ 30%)
* active residual pockets (positive bleeding on probing; BoP) associated with intrabony defects that were not resolved with non-surgical treatment after 4-6 months of maintenance.
* periodontal lesions with probing depth (PD) > 6 mm and supraalveolar defect (pre-diagnosis clinically (periodontal probe)

Exclusion Criteria:

* systemic disease contraindicating periodontal surgery,
* smokers, and
* third molars or teeth with incorrect
* endodontic or restorative treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
interproximal clinical attachment level gain | 6 MONTHS
  measured from CEJ to base of pocket depth by using periodontal prob

SECONDARY OUTCOMES:
residual pocket depth | 6 MONTHS
  distance from gingival margin to pocket depth by using periodontal prob

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University- Russian University in Egypt, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Non-Incised Papilla Flap